CLINICAL TRIAL: NCT01856595
Title: A Phase 1, Placebo-controlled Trial To Assess The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Multiple Escalating Oral Doses Of Pf-06291874 In Adults With Type 2 Diabetes Mellitus
Brief Title: PF-06291874 Multiple Ascending Dose Study In Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B4801003
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — PF-06291874

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-06291874 (Experimental)
  Interventions: Drug: PF-06291874
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06291874 — The dosing schedule is 5, 15, 50, 100 and 150 mg QD for 14 days for the first 5 cohorts in Part A. The dosing schedule for the first cohort in Part B is 15 mg QD for 14 days and 30 mg QD for 28 days
  Arms: PF-06291874
Drug: Placebo — Placebo tablets will be administered QD in each of the cohorts for 14 days (Part A cohorts 1- 5 and Part B cohort 1) or 28 days (Part B cohort 2).
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple ascending doses of PF-06291874 in Type 2 Diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and female subjects of non-childbearing potential between the ages of 18 and 70 years, inclusive of age at the time of the screening visit.

Female subjects of non-childbearing potential must meet at least one of the following criteria:

1. Achieved postmenopausal status, defined as: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum FSH level within the laboratory's reference range for postmenopausal females;
2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
3. Have medically confirmed ovarian failure.
4. All other female subjects (including females with tubal ligations and females that do NOT have a documented hysterectomy, bilateral oophorectomy and/or ovarian failure) will be considered to be of childbearing potential.

   * Body Mass Index (BMI) of 18.0 to 45.0 kg/m2; and a total body weight >50 kg (110 lbs).
   * An informed consent document signed and dated by the subject.
   * Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

PART A ONLY: Subjects treated with metformin monotherapy for at least 3 months at the time of the screening visit; and have been on a stable dose of metformin for at least 6 weeks prior to the first dose of study drug on Day 1. Subjects must be taking a minimum total metformin daily dose of least 1000 mg. Subjects treated with a dipeptidyl peptidase-4 inhibitor (DPP-4i), a sulfonylurea or a sodium-glucose cotransporter-2 inhibitor (SGLT-2i) in combination with metformin may be eligible if washed off the DPP-4i, sulfonylurea or SGLT-2i for a minimum of 4 weeks prior to dosing. Subjects being washed off a DPP-4i, sulfonylurea or SGLT-2i will still need to meet the fasting glucose requirements as defined in the Inclusion Criteria.

PART B ONLY: Subjects treated with metformin plus a sulfonylurea for at least 3 months at the time of the screening visit; and have been on a stable dose of metformin and a sulfonylurea for at least 6 weeks prior to first dose of study drug on Day 1. Subjects must be taking a minimum total metformin daily dose of least 1000 mg and a total daily dose of sulfonylurea that is at least the minimum recommended starting dose found in the product label. Subjects treated with a DPP-4i or SGLT-2i in combination with metformin and a sulfonylurea may be eligible if washed off the DPP-4i or SGLT-2i for a minimum of 4 weeks before dosing.

Exclusion Criteria:

* History of Type 1 diabetes mellitus or secondary forms of diabetes.
* One or more self-reported hypoglycemic episodes of severe intensity within 3 months of screening; or two or more self-reported hypoglycemic episodes of severe intensity within the last 6 months.
* Recent [ie, within six (6) months prior to screening] evidence or medical history of unstable concurrent disease such as: clinically significant hematological, endocrine,pulmonary, gastrointestinal (including severe gastroparesis), cardiovascular, hepatic, psychiatric, neurologic, or clinically significant allergic disease (excluding treated and untreated seasonal allergies at time of dosing). Subjects who have chronic conditions other than T2DM (for example, hypercholesterolemia or hypertension) but are controlled by either diet or stable (for the last 4 weeks prior to screening) doses of medications may be included as well (for example, a subject with hypercholesterolemia on appropriate treatment is eligible).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2013-05-13 (Actual); Primary Completion 2014-01-10 (Actual); Study Completion 2014-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Anaheim Clinical Trials, Anaheim, California
  - Profil Institute for Clinical Research, Inc., Chula Vista, California
  - MRA Clinical Research, LLC, South Miami, Florida

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4801003&StudyName=PF-06291874%20Multiple%20Ascending%20Dose%20Study%20In%20Type%202%20Diabetes%20Mellitus%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Placebo; Part B: Placebo: Participants received placebo matched to PF-06291874 orally once daily for 14 or 28 days
- Part A: PF-06291874 5 mg: Participants received PF-06291874 5 milligram (mg) orally once daily for 14 days
- Part A: PF-06291874 15 mg; Part B: PF-06291874 15 mg: Participants received PF-06291874 15 mg orally once daily for 14 days
- Part A: PF-06291874 50 mg: Participants received PF-06291874 50 mg orally once daily for 14 days
- Part A: PF-06291874 100 mg: Participants received PF-06291874 100 mg orally once daily for 28 days
- Part A: PF-06291874 150 mg: Participants received PF-06291874 150 mg orally once daily for 14 days
- Part B: PF-06291874 30 mg: Participants received PF-06291874 30 mg orally once daily for 28 days
Period: Overall Study
Arm/Group | Part A: Placebo | Part A: PF-06291874 5 mg | Part A: PF-06291874 15 mg | Part A: PF-06291874 50 mg | Part A: PF-06291874 100 mg | Part A: PF-06291874 150 mg | Part B: Placebo | Part B: PF-06291874 15 mg | Part B: PF-06291874 30 mg
Started | 18 | 12 | 12 | 12 | 14 | 12 | 13 | 10 | 14
Completed | 18 | 11 | 12 | 12 | 14 | 12 | 12 | 10 | 14
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: PF-06291874 5 mg | Part A: PF-06291874 15 mg | Part A: PF-06291874 50 mg | Part A: PF-06291874 100 mg | Part A: PF-06291874 150 mg | Part B: Placebo | Part B: PF-06291874 15 mg | Part B: PF-06291874 30 mg | Total
Number analyzed (Participants) | 18 | 12 | 12 | 12 | 14 | 12 | 13 | 10 | 14 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (5.1) | 58.9 (5) | 53.8 (5.9) | 56.2 (7.7) | 54 (10.8) | 56.1 (6.7) | 56.3 (7.6) | 54.2 (8.7) | 55 (10) | 56.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 9 | 4 | 7 | 3 | 4 | 3 | 2 | 47
  Male | 10 | 5 | 3 | 8 | 7 | 9 | 9 | 7 | 12 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Had Protocol-Defined Total Hypoglycemic Adverse Event (HAE) - Part A
Description: A hypoglycemic event (HAE) was identified by characteristic symptoms or blood glucose levels. Hypoglycaemia was assessed and reported in several categories: severe hypoglycaemia, documented symptomatic hypoglycaemia, asymptomatic hypoglycaemia, and probable hypoglycaemia.
Time Frame: Day 1 up to 7-11 days after last dose of study drug
Population: The Safety Analysis Set was defined as all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- Placebo: Participants received placebo orally once daily for 14 or 28 days
- PF-06291874 5 mg: Participants received PF-06291874 5 mg orally once daily for 14 days
- PF-06291874 15 mg: Participants received PF-06291874 15 mg orally once daily for 14 days
- PF-06291874 50 mg: Participants received PF-06291874 50 mg orally once daily for 14 days
- PF-06291874 100 mg: Participants received PF-06291874 100 mg orally once daily for 28 days
- PF-06291874 150 mg: Participants received PF-06291874 150 mg orally once daily for 14 days
Arm/Group | Placebo | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 18 | 12 | 12 | 12 | 14 | 12
participants | 2 | 2 | 1 | 1 | 1 | 2

2. Primary Outcome: Number of Participants Had Protocol-Defined Total Hypoglycemic Adverse Event (HAE) - Part B
Description: as for outcome 1
Time Frame: Day 1 up to 7-11 days after last dose of study drug
Population: The Safety Analysis Set was defined as all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- PF-06291874 30 mg: Participants received PF-06291874 30 mg orally once daily for 28 days
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 30 mg
Number analyzed (Participants) | 13 | 10 | 14
participants | 7 | 4 | 13

3. Primary Outcome: Number of Participants With Electrocardiograms (ECGs) Data Met Criteria of Potential Clinical Concern - Part A
Description: ECG criteria of potential clinical concern were 1), PR interval: greater than or equal to (>=)300 milliseconds (msec); >=25 percent (%) increase when baselinegreater than (>)200 msec; or increase >=50% when baseline less than or equal to (<=)200 msec; 2), QRS interval: >=140 msec; >=50% increase from baseline; 3), QT interval: >=500 msec, QTc interval using cridericia's formula (QTcF interval): absolute value >=450 - <480 msec, >=480-<500 msec, >500 msec; absolute change 30 - <60, >=60 msec.
Time Frame: Predose (0),4,6,8,12,24 hours on Days 1 and 14; 8 hours post dose on Days 3,7,11 for all Cohorts ; predose on Day 17 for Cohorts 1- 4A and 1B; predose on Days 21 and 28 for Cohorts 5A and 2B.
Population: The Safety Analysis Set was defined as all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 18 | 12 | 12 | 12 | 14 | 12
participants
  PR interval >=300 msec | 0 | 0 | 0 | 0 | 0 | 0
  QRS interval >=140 msec | 0 | 0 | 0 | 0 | 0 | 0
  QT interval >=500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval 450-480 msec | 1 | 0 | 1 | 0 | 0 | 1
  QTcF interval 480-500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval >=500 msec | 0 | 0 | 0 | 0 | 0 | 0
  PR interval increase ≥25%/50% | 0 | 0 | 0 | 1 | 0 | 0
  QRS interval increase >=50% | 0 | 0 | 0 | 0 | 0 | 0
  QTcF increase 30-60 msec | 0 | 0 | 1 | 1 | 0 | 0
  QTcF increase >=60 msec | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With ECGs Data Met Criteria of Potential Clinical Concern - Part B
Description: ECG criteria of potential clinical concern were 1), PR interval: >=300 msec; >=25% increase when baseline >200 msec; or increase >=50% when baseline <=200 msec; 2), QRS interval: >=140 msec; >=50% increase from baseline; 3), QT interval: >=500 msec, QTcF interval: absolute value >=450 - <480 msec, >=480-<500 msec, >500 msec; absolute change 30 - <60, >=60 msec.
Time Frame: as for outcome 3
Population: The Safety Analysis Set was defined as all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 30 mg
Number analyzed (Participants) | 13 | 10 | 14
participants
  PR interval >=300 msec | 0 | 0 | 0
  QRS interval >=140 msec | 0 | 0 | 0
  QT interval >=500 msec | 0 | 0 | 0
  QTcF interval 450-480 msec | 1 | 1 | 2
  QTcF interval 480-500 msec | 0 | 0 | 0
  QTcF interval >=500 msec | 0 | 0 | 0
  PR interval increase ≥25%/50% | 0 | 0 | 0
  QRS interval increase >=50% | 0 | 0 | 0
  QTcF increase 30-60 msec | 1 | 0 | 1
  QTcF increase >=60 msec | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Vital Signs Data Met Criteria of Potential Clinical Concern - Part A
Description: Vital signs included blood pressure (BP; supine, sitting and standing) and pulse rate. Vital signs criteria of potential clinical concern were 1), BP: systolic BP (SBP) greater than or equal to (>=) 30 millimeters of mercury (mm Hg) change from grand baseline in same posture, systolic less than (<) 90 mm Hg; diastolic BP (DBP) >=20 mm Hg change from grand baseline in same posture, diastolic <50 mm Hg; 2), pulse rate (supine): <40 or greater than (>) 120 beats per minute (bpm).
Time Frame: as for outcome 3
Population: The Safety Analysis Set was defined as all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 18 | 12 | 12 | 12 | 14 | 12
participants
  Supine SBP <90 mm Hg | 1 | 0 | 0 | 0 | 1 | 0
  Supine DBP <50 mm Hg | 0 | 0 | 0 | 0 | 0 | 0
  Supine pulse rate <40 bpm | 0 | 0 | 0 | 0 | 0 | 0
  Increase:supine SBP≥30 mm Hg | 0 | 0 | 1 | 0 | 0 | 0
  Increase:supine DBP≥20 mm Hg | 3 | 0 | 0 | 0 | 7 | 2
  Decrease:supine SBP≥30 mm Hg | 2 | 1 | 0 | 0 | 0 | 0
  Decrease:supine DBP≥20 mm Hg | 1 | 3 | 1 | 2 | 0 | 0
  Supine pulse rate >120 bpm | 3 | 2 | 1 | 3 | 1 | 0

6. Primary Outcome: Number of Participants With Vital Signs Data Met Criteria of Potential Clinical Concern - Part B
Description: Vital signs included blood pressure (BP; supine, sitting and standing) and pulse rate. Vital signs criteria of potential clinical concern were 1), BP: SBP >= 30 mm Hg change from grand baseline in same posture, SBP < 90 mm Hg; DBP >=20 mm Hg change from grand baseline in same posture, DBP<50 mm Hg; 2), pulse rate (supine): <40 or > 120 bpm.
Time Frame: as for outcome 3
Population: The Safety Analysis Set was defined as all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 30 mg
Number analyzed (Participants) | 13 | 10 | 14
participants
  Supine SBP <90 mm Hg | 1 | 0 | 0
  Supine DBP <50 mm Hg | 0 | 0 | 1
  Supine pulse rate <40 bpm | 0 | 0 | 0
  Increase:supine SBP≥30 mm Hg | 0 | 0 | 0
  Decrease:supine SBP≥30 mm Hg | 3 | 0 | 2
  Decrease:supine DBP≥20 mm Hg | 0 | 1 | 0
  Supine pulse rate >120 bpm | 0 | 1 | 0
  Increase:supine DBP≥20 mm Hg | 2 | 0 | 3

7. Primary Outcome: Number of Participants With Any Abnormal Laboratory Test Results - Part A
Description: The laboratory test included: hematology (hemoglobin, hematocrit, red blood cell count, MCV, MCH, MCHC, platelets, white blood cell count, absolute lymphocytes, absolute total neutrophils, absolute basophils, absolute eosinophils and absolute monocytes), coagulation (PPT, prothrombin), liver function(total bilirubin, AST, ALT, alkaline phosphatase, total protein and albumin), renal function (blood urea nitrogen, creatinine, uric acid), Lipids (cholesterol, HDL cholesterol, LDL cholesterol, triglycerides), Electrolytes (sodium, potassium, chloride, calcium, venous bicarbonate), clinical chemistry (glucose, glycosylated, hemoglobin, amylase, lipase), urinalysis dipstick (urine PH, urine glucose, urine ketones, urine protein, urine urobilinogen, urine bilirubin, urine nitrite, urine leukocyte, esterase), urinalysis microscopy (urine RBC, urine WBC, urine bacteria). Laboratory abnormality was determined by the investigator based on pre-defined criteria.
Time Frame: Predose on Days 0,3,7,11 for all cohorts and 14 and 17 for Cohorts 1- 4A and 1B, and pre-dose on Days 21 and 28 for Cohorts 5A and 2B.
Population: The Safety Analysis Set was defined as all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 18 | 12 | 12 | 12 | 14 | 12
participants | 17 | 10 | 11 | 12 | 13 | 8

8. Primary Outcome: Number of Participants With Any Abnormal Laboratory Test Results - Part B
Description: as for outcome 7
Time Frame: as for outcome 7
Population: The Safety Analysis Set was defined as all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-06291874 5 mg | PF-06291874 30 mg | Placebo
Number analyzed (Participants) | 10 | 14 | 13
participants | 8 | 12 | 11

9. Primary Outcome: Single Dose Maximum Plasma Concentration (Cmax) for PF-06291874 - Part A
Description: Cmax was maximum plasma concentration. Blood samples (3 mL) to provide a minimum of approximately 1.2 mL plasma for pharmacokinetic (PK) analysis were collected at 0, 2, 4, 6, 8, 12, 19 and 24 hours post dose.
Time Frame: 0 hour (pre-dose), 2, 4, 6, 8, 12, 19, 24 hours post-dose on Day 1
Population: This PK Parameter Analysis Set was defined as all participants randomized and treated who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 12 | 12 | 12 | 14 | 12
nanograms per milliliter (ng/mL) | 137.0 (17) | 427.1 (22) | 1308 (26) | 2582 (19) | 3288 (32)

10. Primary Outcome: Single Dose Normalized Cmax (Cmax[dn]) for PF-06291874 - Part A
Description: Cmax (dn) was dose normalized maximum plasma concentration. Blood samples (3 mL) to provide a minimum of approximately 1.2 mL plasma for pharmacokinetic (PK) analysis were collected at 0, 2, 4, 6, 8, 12, 19 and 24 hours post dose.
Time Frame: 0 hour (pre-dose), 2, 4, 6, 8, 12, 19, 24 hours post-dose on Day 1
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 12 | 12 | 12 | 14 | 12
ng/mL/mg | 27.40 (17) | 28.46 (22) | 26.15 (26) | 25.82 (19) | 21.90 (32)

11. Primary Outcome: Single Dose Cmax for PF-06291874 - Part B
Description: Cmax was maximum plasma concentration. Blood samples (3 mL) to provide a minimum of approximately 1.2 mL plasma for PK analysis were collected at 0, 2, 4, 6, 8, 12, 19 and 24 hours post dose.
Time Frame: 0 hour (pre-dose), 2, 4, 6, 8, 12, 19, 24 hours post-dose on Day 1
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06291874 15 mg | PF-06291874 30 mg
Number analyzed (Participants) | 10 | 14
ng/mL | 373.6 (16) | 687.6 (34)

12. Primary Outcome: Single Dose Normalized Cmax (Cmax[dn]) for PF-06291874 - Part B
Description: Cmax (dn) was dose normalized maximum plasma concentration. Blood samples (3 mL) to provide a minimum of approximately 1.2 mL plasma for PK analysis were collected at 0, 2, 4, 6, 8, 12, 19 and 24 hours post dose
Time Frame: 0 hour (pre-dose), 2, 4, 6, 8, 12, 19, 24 hours post-dose on Day 1
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | PF-06291874 15 mg | PF-06291874 30 mg
Number analyzed (Participants) | 10 | 14
ng/mL/mg | 24.90 (16) | 22.92 (34)

13. Primary Outcome: Single Dose Time at Which Cmax Occurred (Tmax) for PF-06291874 - Part A
Description: Tmax was time at which Cmax occurred. Blood samples (3 mL) to provide a minimum of approximately 1.2 mL plasma for PK analysis were collected at 0, 2, 4, 6, 8, 12, 19, 24 hours post dose.
Time Frame: 0 hour (pre-dose), 2, 4, 6, 8, 12, 19, 24 hours post-dose on Day 1
Population: as for outcome 9
Measure: Median (Full Range); unit: hr
Arm/Group | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 12 | 12 | 12 | 14 | 12
hr | 6.00 (17) [2.00 to 8.03] | 5.00 (22) [4.00 to 12.0] | 6.00 (26) [2.00 to 8.02] | 6.07 (19) [4.00 to 8.00] | 4.00 (32) [2.00 to 8.00]

14. Primary Outcome: Single Dose Tmax for PF-06291874 - Part B
Description: as for outcome 13
Time Frame: 0 hour (pre-dose), 2, 4, 6, 8, 12, 19, 24 hours post-dose on Day 1
Population: as for outcome 9
Measure: Median (Full Range); unit: hr
Arm/Group | PF-06291874 15 mg | PF-06291874 30 mg
Number analyzed (Participants) | 10 | 14
hr | 6.02 (16) [4.00 to 12.0] | 6.00 (34) [2.00 to 12.0]

15. Primary Outcome: Single Dose AUCtau (Area Under the Concentration-time Profile From Time Zero to Time Tau, the Dosing Interval, Where Tau = 24 Hours) for PF-06291874 - Part A
Description: AUCtau was area under the concentration-time profile from time zero to time tau, the dosing interval, where tau = 24 hours. Blood samples (3 mL) to provide a minimum of approximately 1.2 mL plasma for PK analysis were collected at 0, 2, 4, 6, 8, 12, 19, 24 hours post dose.
Time Frame: 0 hour (pre-dose), 2, 4, 6, 8, 12, 19, 24 hours post-dose on Day 1
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hr/mL
Arm/Group | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 12 | 12 | 12 | 14 | 12
ng.hr/mL | 2181 (27) [2.00 to 8.03] | 6821 (20) [4.00 to 12.0] | 20650 (27) [2.00 to 8.02] | 43040 (20) [4.00 to 8.00] | 51860 (34) [2.00 to 8.00]

16. Primary Outcome: Single Dose AUCtau for PF-06291874 - Part B
Description: as for outcome 15
Time Frame: 0 hour (pre-dose), 2, 4, 6, 8, 12, 19, 24 hours post-dose on Day 1
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hr/mL
Arm/Group | PF-06291874 15 mg | PF-06291874 30 mg
Number analyzed (Participants) | 10 | 14
ng.hr/mL | 6486 (14) [4.00 to 12.0] | 11280 (35) [2.00 to 12.0]

17. Primary Outcome: Multiple Dose Cmax for PF-06291874 - Part A
Description: Cmax was maximum plasma concentration. Blood samples (3 mL) to provide a minimum of approximately 1.2 mL plasma for PK analysis were collected at 0, 2, 4, 6, 8, 12, 19, 24 hours post dose.
Time Frame: Predose (0), 2, 4, 6, 8, 12, 19, 24 hours post dose on Day 14
Population: This PK Parameter Analysis Set was defined as all participants randomized and treated who had at least 1 of the PK parameters of interest. The number of participants analyzed was the number of participants contributing to the summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 11 | 12 | 12 | 14 | 12
ng/mL | 213.4 (27) | 669.1 (17) | 2220 (31) | 4362 (30) | 5957 (29)

18. Primary Outcome: Multiple Dose Cmax for PF-06291874 - Part B
Description: as for outcome 17
Time Frame: Predose (0), 2, 4, 6, 8, 12, 19, 24 hours post dose on Day 14
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06291874 15 mg | PF-06291874 30 mg
Number analyzed (Participants) | 10 | 14
ng/mL | 663.1 (19) | 1108 (26)

19. Primary Outcome: Multiple Dose Tmax for PF-06291874 - Part A
Description: as for outcome 13
Time Frame: Predose (0), 2, 4, 6, 8, 12, 19, 24 hours post dose on Day 14
Population: as for outcome 17
Measure: Median (Full Range); unit: hour
Arm/Group | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 11 | 12 | 12 | 14 | 12
hour | 5.98 [4.00 to 12.0] | 5.00 [4.00 to 8.00] | 4.02 [2.02 to 6.00] | 6.00 [2.02 to 12.0] | 5.00 [1.98 to 12.2]

20. Primary Outcome: Multiple Dose Tmax for PF-06291874 - Part B
Description: as for outcome 13
Time Frame: Predose (0), 2, 4, 6, 8, 12, 19, 24 hours post dose on Day 14
Population: as for outcome 9
Measure: Median (Full Range); unit: hr
Arm/Group | PF-06291874 15 mg | PF-06291874 30 mg
Number analyzed (Participants) | 10 | 14
hr | 4.00 (19) [1.95 to 6.00] | 6.00 (26) [2.02 to 12.0]

21. Primary Outcome: Multiple Dose AUCtau for PF-06291874 - Part A
Description: as for outcome 15
Time Frame: Predose (0), 2, 4, 6, 8, 12, 19, 24 hours post dose on Day 14
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hr/mL
Arm/Group | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 11 | 12 | 12 | 14 | 12
ng.hr/mL | 3800 (42) [2.00 to 8.03] | 11760 (19) [4.00 to 12.0] | 39560 (30) [2.00 to 8.02] | 79550 (32) [4.00 to 8.00] | 105400 (37) [2.00 to 8.00]

22. Primary Outcome: Multiple Dose AUCtau for PF-06291874 - Part B
Description: as for outcome 15
Time Frame: Predose (0), 2, 4, 6, 8, 12, 19, 24 hours post dose on Day 14
Population: This PK Parameter Analysis Set was defined as all participants randomized and treated who have at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hr/mL
Arm/Group | PF-06291874 15 mg | PF-06291874 30 mg
Number analyzed (Participants) | 10 | 14
ng.hr/mL | 11530 (23) [4.00 to 12.0] | 19270 (34) [2.00 to 12.0]

23. Primary Outcome: Multiple Dose Half Life for PF-06291874
Description: Plasma half-life was the time measured for the plasma concentration to decrease by one half. Blood samples (3 mL) to provide a minimum of approximately 1.2 mL plasma for PK analysis were collected at 0, 2, 4, 6, 8, 12, 19, 24 hours post dose.
Time Frame: Predose (0), 2, 4, 6, 8, 12, 19, 24 hours post dose on Day 14
Population: This PK Parameter Analysis Set was defined as all participants randomized and treated who have at least 1 of the PK parameters of interest. The number of participants analyzed was the number of participants contributing to the summary statistics. This parameter was not calculated for group: 100 mg Part A, 30 mg Part B.
Measure: Mean (Standard Deviation); unit: hr
Groups:
- PF-06291874 15 mg - Part B: Participants received PF-06291874 15 mg orally once daily for 14 days
Arm/Group | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 150 mg | PF-06291874 15 mg - Part B
Number analyzed (Participants) | 11 | 12 | 11 | 12 | 10
hr | 20.96 (5.6029) [2.00 to 8.03] | 19.68 (4.2407) [4.00 to 12.0] | 22.24 (3.2605) [2.00 to 8.02] | 20.83 (4.1134) [2.00 to 8.00] | 22.74 (3.4699)

24. Primary Outcome: Multiple Dose Cmin (Lowest Plasma Concentration Observed During the Dosing Interval) for PF-06291874 - Part A
Description: Cmin was the lowest plasma concentration observed during the dosing interval. Blood samples (3 mL) to provide a minimum of approximately 1.2 mL plasma for PK analysis were collected at 0, 2, 4, 6, 8, 12, 19, 24 hours post dose.
Time Frame: Predose (0), 2, 4, 6, 8, 12, 19, 24 hours post dose on Day 14
Population: This PK Parameter Analysis Set was defined as all participants randomized and treated who have at least 1 of the PK parameters of interest. The number of participants analyzed was the number of participants contributing to the summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 11 | 12 | 12 | 14 | 12
ng/mL | 117.8 (58) | 350.5 (28) | 1132 (38) | 1747 (178) | 3096 (47)

25. Primary Outcome: Multiple Dose Cmin for PF-06291874 - Part B
Description: as for outcome 24
Time Frame: Predose (0), 2, 4, 6, 8, 12, 19, 24 hours post dose on Day 14
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06291874 15 mg | PF-06291874 30 mg
Number analyzed (Participants) | 10 | 14
ng/mL | 339.5 (32) | 411.5 (217)

26. Primary Outcome: Multiple Dose Apparent Clearance (CL/F) for PF-06291874 - Part A
Description: CL/F was multiple dose apparent clearance. The 24-hour urine samples for PK analysis were collected on Day 14 over 2 collection periods (0-6 hours and 6-24 hours).
Time Frame: on Day 14 over 2 collection periods (0-6 hours and 6-24 hours).
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 11 | 12 | 12 | 14 | 12
L/hr | 1.315 (42) | 1.275 (19) | 1.264 (30) | 1.258 (32) | 1.422 (37)

27. Primary Outcome: Multiple Dose CL/F for PF-06291874 - Part B
Description: as for outcome 26
Time Frame: on Day 14 over 2 collection periods (0-6 hours and 6-24 hours).
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-06291874 15 mg | PF-06291874 30 mg
Number analyzed (Participants) | 10 | 14
L/hr | 1.300 (23) | 1.555 (34)

28. Primary Outcome: Multiple Dose Apparent Volume of Distribution (Vz/F) for PF-06291874- Part A and Part B
Description: Vz/F was apparent volume of distribution. Blood samples (3 mL) to provide a minimum of approximately 1.2 mL plasma for PK analysis were collected at 0, 2, 4, 6, 8, 12, 19, 24 hours post dose.
Time Frame: Predose (0), 2, 4, 6, 8, 12, 19, 24 hours post dose on Day 14
Population: This PK Parameter Analysis Set was defined as all participants randomized and treated who have at least 1 of the PK parameters of interest. This parameter was not calculated for treatment groups with only 24-hour sampling on Day 14(A: 100 mg and B: 30 mg), since the terminal phase was not well characterized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 150 mg | PF-06291874 15 mg - Part B
Number analyzed (Participants) | 11 | 12 | 11 | 12 | 10
L | 38.37 (20) | 35.54 (21) | 40.47 (25) | 41.88 (29) | 42.20 (14)

29. Primary Outcome: Multiple Dose Observed Accumulation Ratio (Rac) for PF-06291874 - Part A
Description: Rac was observed accumulation ratio. Blood samples (3 mL) to provide a minimum of approximately 1.2 mL plasma for PK analysis were collected at 0, 2, 4, 6, 8, 12, 19, 24 hours post dose.
Time Frame: Predose (0), 2, 4, 6, 8, 12, 19, 24 hours post dose on Day 14
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 11 | 12 | 12 | 14 | 12
ratio | 1.766 (38) | 1.724 (17) | 1.915 (17) | 1.847 (22) | 2.032 (16)

30. Primary Outcome: Multiple Dose Rac for PF-06291874 - Part B
Description: as for outcome 29
Time Frame: Predose (0), 2, 4, 6, 8, 12, 19, 24 hours post dose on Day 14
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-06291874 15 mg | PF-06291874 30 mg
Number analyzed (Participants) | 10 | 14
ratio | 1.780 (17) | 1.709 (22)

31. Primary Outcome: Multiple Dose Rac for Cmax (Rac,Cmax) for PF-06291874 - Part A
Description: Rac,cmax was observed accumulation ratio for Cmax. Blood samples (3 mL) to provide a minimum of approximately 1.2 mL plasma for PK analysis were collected at 0, 2, 4, 6, 8, 12, 19, 24 hours post dose.
Time Frame: Predose (0), 2, 4, 6, 8, 12, 19, 24 hours post dose on Day 14
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 11 | 12 | 12 | 14 | 12
ratio | 1.575 (26) | 1.567 (23) | 1.698 (19) | 1.690 (25) | 1.812 (18)

32. Primary Outcome: Multiple Dose Rac,Cmax for PF-06291874 - Part B
Description: as for outcome 31
Time Frame: Predose (0), 2, 4, 6, 8, 12, 19, 24 hours post dose on Day 14
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-06291874 15 mg | PF-06291874 30 mg
Number analyzed (Participants) | 10 | 14
ratio | 1.775 (22) | 1.610 (16)

33. Primary Outcome: Multiple Dose Percent of Cumulative Amount of Drug Recovered Unchanged in Urine Over the Dosing Interval τ(Aetau%) for PF-06291874
Description: Aetau% was percent of cumulative amount of drug recovered unchanged in urine over the dosing interval τ. The 24-hour urine samples for PK analysis were collected on Day 14 over 2 collection periods (0-6 hours and 6-24 hours).
Time Frame: on Day 14 over 2 collection periods (0-6 hours and 6-24 hours).
Population: This PK Parameter Analysis Set was defined as all participants randomized and treated who have at least 1 of the PK parameters of interest. For treatment groups with dose< 50 mg, all urine concentrations were below the lower limit of quantification (<50.0 ng/mL) and hence no urine parameter was calculated including Aetau%.
Measure: Median (Full Range); unit: percentage of dose
Arm/Group | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 11 | 14 | 12
percentage of dose | 0.0000 (19) [0.000 to 0.0686] | 0.0000 (25) [0.000 to 0.232] | 0.0000 (18) [0.000 to 0.256]

34. Primary Outcome: Multiple Dose Renal Clearance (CLr) for PF-06291874
Description: CLr was renal clearance. The 24 hour urine samples for PK analysis were collected on Day 14 over 2 collection periods (0-6 hours and 6-24 hours)
Time Frame: on Day 14 over 2 collection periods (0-6 hours and 6-24 hours).
Population: This PK Parameter Analysis Set was defined as all participants randomized and treated who have at least 1 of the PK parameters of interest. For treatment groups with dose< 50 mg, all urine concentrations were below the lower limit of quantification (<50.0 ng/mL) and hence no urine parameter was calculated including CLr.
Measure: Median (Full Range); unit: mL/hr
Arm/Group | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 11 | 14 | 12
mL/hr | 0.0000 (19) [0.000 to 0.441] | 0.0000 (25) [0.000 to 2.25] | 0.0000 (18) [0.000 to 2.49]

35. Primary Outcome: Changes From Baseline for Mean Daily Glucose (mg/dL) on Day 14 (AUC Approach) - Part A
Description: A MMTT was administered on Days -1 and 14 for all cohorts. Blood samples for analysis of glucose were collected at nominal time 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 10, 12, 15, 19 and 24 hours on Days -1 and 14 for all cohorts. MDG was computed by AUC24/24 hours of the glucose values measured.
Time Frame: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 10, 12, 15, 19 and 24 hours on Days -1 and 14 for all cohorts, and on Day 28 for PF-06291874 100 mg Part A and PF-06291874 30 mg Part B.
Population: All subjects administered PF-06291874 or placebo were included in PD analysis. Placebo subjects within each cohort in Part A or B were pooled into a single placebo group for the inpatient portion of the study. Data collected from placebo subjects during the outpatient portion of study (Day 28) were also pooled separately for Parts A and B.
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 18 | 11 | 12 | 12 | 14 | 12
mg/dL | -11.54 (58) [-20.26 to -2.81] | -14.31 (28) [-25.47 to -3.16] | -33.18 (38) [-43.96 to -22.40] | -38.13 (178) [-48.83 to -27.43] | -43.86 (47) [-53.89 to -33.84] | -53.92 [-64.72 to -43.13]
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 5 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.7457, ANCOVA — Two-sided p-values are from analysis of Covariance (ANCOVA) model with treatment as a factor and baseline value as a covariate. P-values are not adjusted for multiple comparisons; Least Square Mean Difference (Net) = -2.77, 90% CI 2-sided [-16.93 to 11.38], Standard Error of Mean 8.532
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 15 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.0108, ANCOVA — [p-value comment as in outcome 35, analysis 1]; Least Square Mean Difference (Net) = -21.64, 90% CI 2-sided [-35.47 to -7.81], Standard Error of Mean 8.334
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 15 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.0018, ANCOVA — [p-value comment as in outcome 35, analysis 1]; Least Square Mean Difference (Net) = -26.59, 90% CI 2-sided [-40.38 to -12.80], Standard Error of Mean 8.309
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 35, analysis 1]; Least Square Mean Difference (Net) = -32.33, 90% CI 2-sided [-45.66 to -18.99], Standard Error of Mean 8.038
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 150 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 35, analysis 1]; Least Square Mean Difference (Net) = -42.39, 90% CI 2-sided [-56.23 to -28.55], Standard Error of Mean 8.340

36. Primary Outcome: Changes From Baseline for Mean Daily Glucose (mg/dL) on Day 14 (AUC Approach) - Part B
Description: as for outcome 35
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Least Squares Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | PF-06291874 15 mg | PF-06291874 30 mg | Placebo
Number analyzed (Participants) | 10 | 14 | 6
ng/mL | -20.85 (32) [-32.56 to -9.15] | -50.65 (217) [-60.58 to -40.71] | -31.32 [-42.12 to -20.52]
Statistical Analysis 1: Comparison: PF-06291874 15 mg vs Placebo; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.2790, ANCOVA — Two-sided p-values are from ANCOVA model with treatment as a factor and baseline value as a covariate. P-values are not adjusted for multiple comparisons; Least Square Mean Difference (Net) = 10.47, 90% CI 2-sided [-5.50 to 26.43], Standard Error of Mean 9.621
Statistical Analysis 2: Comparison: PF-06291874 30 mg vs Placebo; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.0299, ANCOVA — [p-value comment as in outcome 36, analysis 1]; Least Square Mean Difference (Net) = -19.33, 90% CI [-33.89 to -4.76], Standard Error of Mean 8.777

37. Primary Outcome: Changes From Baseline for Mean Daily Glucose (mg/dL) on Day 28 (AUC Approach)
Description: A MMTT was administered on Days -1 for all cohorts, and on Day 28 for PF-06291874 100 mg Part A and PF-06291874 30 mg Part B. Blood samples for analysis of glucose were collected at nominal time 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 10, 12, 15, 19 and 24 hours on Days -1 and 14 for all cohorts, and on Day 28 for PF-06291874 100 mg Part A and PF-06291874 30 mg Part B. MDG was computed by AUC24/24 hours of the glucose values measured.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Groups:
- Placebo - Part B: Participants received placebo orally once daily for 14 or 28 days
- PF-06291874 30 mg - Part B: Participants received PF-06291874 30 mg orally once daily for 14 days
Arm/Group | Placebo | PF-06291874 100 mg | Placebo - Part B | PF-06291874 30 mg - Part B
Number analyzed (Participants) | 6 | 14 | 7 | 13
mg/dL | -6.99 (58) [-17.73 to 3.75] | -36.42 (28) [-43.44 to -29.39] | -30.10 (38) [-40.05 to -20.16] | -42.00 (178) [-49.29 to -34.70]
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.0005, ANCOVA — [p-value comment as in outcome 35, analysis 1]; Least Square Mean Difference (Net) = -29.43, 90% CI 2-sided [-42.28 to -16.57], Standard Error of Mean 7.609
Statistical Analysis 2: Comparison: Placebo - Part B vs PF-06291874 30 mg - Part B; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.1133, ANCOVA — [p-value comment as in outcome 35, analysis 1]; Least Square Mean Difference (Net) = -11.89, 90% CI 2-sided [-24.26 to 0.48], Standard Error of Mean 7.321

38. Secondary Outcome: Changes Relative to Baseline (Ratio) of AUC0-4 for Glucose Following MMTT on Day 14 - Part A
Description: Blood samples for analysis of glucose were collected at nominal time 0, 0.25, 0.5, 1, 1.5, 2, 3, and 4 hours on Days -1 and 14 for all cohorts, and on Day 28 for PF-06291874 100 mg Part A and PF-06291874 30 mg Part B. AUC0-4 and natural log transformed AUC0-4 were calculated for each day.
Time Frame: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 10, 12, 15, and 19 hours on Days -1 and 14 for all cohorts, and on Day 28 for PF-06291874 100 mg Part A and PF-06291874 30 mg Part B.
Population: as for outcome 35
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Placebo | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 18 | 11 | 12 | 12 | 14 | 12
ratio | 0.88 [0.82 to 0.94] | 0.87 [0.80 to 0.94] | 0.75 [0.69 to 0.82] | 0.74 [0.69 to 0.81] | 0.72 [0.67 to 0.77] | 0.67 [0.62 to 0.73]
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 5 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.8530, ANCOVA — Two-sided p-values are from analysis of Covariance (ANCOVA) model with treatment as a factor and baseline value as a covariate using the natural log-transformed AUC0-4. P-values are not adjusted for multiple comparisons; Ratio = 0.99, 90% CI 2-sided [0.89 to 1.10], Standard Error of Mean 1.066
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 15 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.0172, ANCOVA — [p-value comment as in outcome 38, analysis 1]; Ratio = 0.86, 90% CI 2-sided [0.77 to 0.95], Standard Error of Mean 1.065
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 50 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.0106, ANCOVA — [p-value comment as in outcome 38, analysis 1]; Ratio = 0.85, 90% CI 2-sided [0.77 to 0.94], Standard Error of Mean 1.064
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.0012, ANCOVA — [p-value comment as in outcome 38, analysis 1]; Ratio = 0.82, 90% CI 2-sided [0.74 to 0.90], Standard Error of Mean 1.062
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 150 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 38, analysis 1]; Ratio = 0.77, 90% CI 2-sided [0.69 to 0.85], Standard Error of Mean 1.065

39. Secondary Outcome: Changes Relative to Baseline (Ratio) of AUC0-4 for Glucose Following MMTT on Day 14 - Part B
Description: as for outcome 38
Time Frame: as for outcome 38
Population: as for outcome 35
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | PF-06291874 15 mg | PF-06291874 30 mg | Placebo
Number analyzed (Participants) | 10 | 14 | 6
ratio | 0.81 (32) [0.74 to 0.89] | 0.74 (217) [0.69 to 0.80] | 0.83 [0.76 to 0.90]
Statistical Analysis 1: Comparison: PF-06291874 15 mg vs Placebo; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.7804, ANCOVA — Two-sided p-values are from analysis of ANCOVA model with treatment as a factor and baseline value as a covariate using the natural log-transformed AUC0-4. P-values are not adjusted for multiple comparisons; Ratio = 0.98, 90% CI 2-sided [0.87 to 1.10], Standard Error of Mean 1.075
Statistical Analysis 2: Comparison: PF-06291874 30 mg vs Placebo; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.0908, ANCOVA — Two-sided p-values are from ANCOVA model with treatment as a factor and baseline value as a covariate using the natural log-transformed AUC0-4. P-values are not adjusted for multiple comparisons; Ratio = 0.88, 90% CI 2-sided [0.77 to 1.00], Standard Error of Mean 1.068

40. Secondary Outcome: Changes Relative to Baseline (Ratio) of AUC0-4 for Glucose Following MMTT on Day 28
Description: as for outcome 38
Time Frame: as for outcome 38
Population: as for outcome 35
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Placebo | PF-06291874 100 mg | Placebo - Part B | PF-06291874 30 mg - Part B
Number analyzed (Participants) | 6 | 14 | 7 | 13
ratio | 1.02 (58) [0.91 to 1.14] | 0.79 (28) [0.73 to 0.85] | 0.89 (38) [0.80 to 0.99] | 0.78 (178) [0.73 to 0.84]
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.0027, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 0.77, 90% CI 2-sided [0.68 to 0.88], Standard Error of Mean 1.083
Statistical Analysis 2: Comparison: Placebo - Part B vs PF-06291874 30 mg - Part B; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.0908, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 0.88, 90% CI 2-sided [0.77 to 1.00], Standard Error of Mean 1.079

41. Secondary Outcome: Percent Changes From Baseline of AUC0-4 for Glucagon Following MMTT on Day 14 - Part A
Description: Blood samples for analysis of insulin, C-peptide, glucagon and glucagon-like peptide 1 (GLP-1) were collected at nominal time 0, 0.25, 0.5, 1, 1.5, 2, 3, 4 hours on Days -1 and 14 for all cohorts, and on Day 28 and follow-up visit for PF-06291874 100 mg Part A and PF-06291874 30 mg Part B. AUC0-4 and natural log transformed AUC0-4 were calculated for each day.
Time Frame: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4 hours on Days -1 and 14 for all cohorts, and on Day 28 and follow-up visit for PF-06291874 100 mg Part A and PF-06291874 30 mg Part B.
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 18 | 11 | 12 | 12 | 14 | 12
Percentage of change | 1.38 (20.396) [0.82 to 0.94] | 12.17 (11.910) [0.80 to 0.94] | 50.45 (37.048) [0.69 to 0.82] | 46.90 (30.179) [0.69 to 0.81] | 142.62 (113.394) [0.67 to 0.77] | 214.32 (118.612) [0.62 to 0.73]

42. Secondary Outcome: Percent Changes From Baseline of AUC0-4 for Glucagon Following MMTT on Day 14 - Part B
Description: as for outcome 41
Time Frame: as for outcome 41
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | PF-06291874 15 mg | PF-06291874 30 mg | Placebo
Number analyzed (Participants) | 12 | 10 | 13
Percentage of change | 33.19 (23.47) [0.74 to 0.89] | 50.35 (24.33) [0.69 to 0.80] | 7.23 (22.59) [0.76 to 0.90]

43. Secondary Outcome: Percent Changes From Baseline of AUC0-4 for Glucagon Following MMTT on Day 28
Description: Blood samples for analysis of insulin, C-peptide, glucagon and GLP-1 were collected at nominal time 0, 0.25, 0.5, 1, 1.5, 2, 3, 4 hours on Days -1 and 14 for all cohorts, and on Day 28 and follow-up visit for PF-06291874 100 mg Part A and PF-06291874 30 mg Part B. AUC0-4 and natural log transformed AUC0-4 were calculated for each day.
Time Frame: as for outcome 41
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo | PF-06291874 100 mg | Placebo - Part B | PF-06291874 30 mg
Number analyzed (Participants) | 6 | 14 | 7 | 13
Percentage of change | 23.04 (52.52) [0.91 to 1.14] | 125.15 (120.82) [0.73 to 0.85] | -1.19 (29.18) [0.80 to 0.99] | 36.49 (45.17) [0.73 to 0.84]

44. Secondary Outcome: Changes Relative to Baseline (Ratio) of AUC0-4 for Insulin Following MMTT on Day 14 - Part A
Description: as for outcome 43
Time Frame: as for outcome 41
Population: All subjects administered PF-06291874 or placebo were included in PD analysis. Placebo subjects within each cohort in Part A or B were pooled into a single placebo group for the inpatient portion of the study. The number of participants analyzed was the number of participants contributing to the summary statistics.
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Placebo | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 18 | 11 | 11 | 11 | 14 | 12
ratio | 1.02 [0.91 to 1.15] | 1.01 [0.86 to 1.17] | 0.95 [0.82 to 1.11] | 0.85 [0.73 to 1.00] | 0.91 [0.80 to 1.04] | 1.00 [0.87 to 1.16]
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 5 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.8723, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 0.98, 90% CI 2-sided [0.81 to 1.19], Standard Error of Mean 1.123
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 15 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.5158, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 0.93, 90% CI 2-sided [0.76 to 1.13], Standard Error of Mean 1.124
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 50 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.1258, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 0.83, 90% CI 2-sided [0.68 to 1.01], Standard Error of Mean 1.126
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.2883, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 0.89, 90% CI 2-sided [0.74 to 1.07], Standard Error of Mean 1.115
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 150 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.8437, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 0.98, 90% CI 2-sided [0.81 to 1.18], Standard Error of Mean 1.120

45. Secondary Outcome: Changes Relative to Baseline (Ratio) of AUC0-4 for Insulin Following MMTT on Day 14 - Part B
Description: as for outcome 43
Time Frame: as for outcome 41
Population: as for outcome 35
Measure: Least Squares Mean (90% Confidence Interval); unit: Ratio
Arm/Group | PF-06291874 15 mg | PF-06291874 30 mg | Placebo
Number analyzed (Participants) | 10 | 14 | 6
Ratio | 1.13 (32) [0.95 to 1.33] | 1.10 (217) [0.95 to 1.28] | 1.01 [0.85 to 1.19]
Statistical Analysis 1: Comparison: PF-06291874 15 mg vs Placebo; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.4405, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 1.12, 90% CI 2-sided [0.88 to 1.42], Standard Error of Mean 1.154
Statistical Analysis 2: Comparison: PF-06291874 30 mg vs Placebo; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.5178, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 1.09, 90% CI 2-sided [0.87 to 1.37], Standard Error of Mean 1.146

46. Secondary Outcome: Changes Relative to Baseline (Ratio) of AUC0-4 for Insulin Following MMTT on Day 28
Description: as for outcome 43
Time Frame: as for outcome 41
Population: as for outcome 35
Measure: Least Squares Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Placebo | PF-06291874 100 mg | Placebo - Part B | PF-06291874 30 mg
Number analyzed (Participants) | 6 | 14 | 7 | 13
Ratio | 1.22 (58) [0.97 to 1.54] | 0.85 (28) [0.73 to 0.99] | 0.77 (38) [0.62 to 0.96] | 0.93 (178) [0.79 to 1.09]
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.0340, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 0.69, 90% CI 2-sided [0.52 to 0.92], Standard Error of Mean 1.181
Statistical Analysis 2: Comparison: Placebo - Part B vs PF-06291874 30 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.2519, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 1.20, 90% CI 2-sided [0.92 to 1.58], Standard Error of Mean 1.173

47. Secondary Outcome: Changes Relative to Baseline (Ratio) of AUC0-4 for C-Peptide Following MMTT on Day 14 - Part A
Description: as for outcome 43
Time Frame: as for outcome 41
Population: as for outcome 35
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Placebo | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 18 | 12 | 12 | 12 | 14 | 12
ratio | 0.96 [0.88 to 1.04] | 1.01 [0.92 to 1.12] | 0.94 [0.85 to 1.04] | 0.89 [0.80 to 0.99] | 0.95 [0.87 to 1.05] | 1.03 [0.94 to 1.14]
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 5 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.4579, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 1.06, 90% CI 2-sided [0.93 to 1.20], Standard Error of Mean 1.079
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 15 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.8144, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 0.98, 90% CI 2-sided [0.87 to 1.11], Standard Error of Mean 1.079
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 50 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.3425, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 0.93, 90% CI 2-sided [0.81 to 1.06], Standard Error of Mean 1.082
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.9670, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 1.00, 90% CI 2-sided [0.88 to 1.13], Standard Error of Mean 1.076
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 150 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.3190, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 1.08, 90% CI 2-sided [0.95 to 1.23], Standard Error of Mean 1.079

48. Secondary Outcome: Changes Relative to Baseline (Ratio) of AUC0-4 for C-Peptide Following MMTT on Day 14 - Part B
Description: as for outcome 43
Time Frame: as for outcome 41
Population: as for outcome 35
Measure: Least Squares Mean (90% Confidence Interval); unit: Ratio
Arm/Group | PF-06291874 15 mg | PF-06291874 30 mg | Placebo
Number analyzed (Participants) | 10 | 14 | 6
Ratio | 1.19 (32) [1.06 to 1.33] | 1.13 (217) [1.03 to 1.24] | 1.05 [0.95 to 1.16]
Statistical Analysis 1: Comparison: PF-06291874 15 mg vs Placebo; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.1617, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 1.14, 90% CI 2-sided [0.98 to 1.32], Standard Error of Mean 1.095
Statistical Analysis 2: Comparison: PF-06291874 30 mg vs Placebo; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.3703, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 1.08, 90% CI 2-sided [0.94 to 1.23], Standard Error of Mean 1.084

49. Secondary Outcome: Changes Relative to Baseline (Ratio) of AUC0-4 for C-Peptide Following MMTT on Day 28
Description: as for outcome 43
Time Frame: as for outcome 41
Population: as for outcome 35
Measure: Least Squares Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Placebo | PF-06291874 100 mg | Placebo - Part B | PF-06291874 30 mg
Number analyzed (Participants) | 6 | 14 | 7 | 14
Ratio | 0.95 (58) [0.81 to 1.11] | 0.91 (28) [0.82 to 1.00] | 0.79 (38) [0.68 to 0.91] | 0.93 (178) [0.84 to 1.03]
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 100 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.6833, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 0.95, 90% CI 2-sided [0.79 to 1.15], Standard Error of Mean 1.119
Statistical Analysis 2: Comparison: Placebo - Part B vs PF-06291874 30 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p = 0.1318, ANCOVA — [p-value comment as in outcome 39, analysis 2]; Ratio = 1.18, 90% CI 2-sided [0.98 to 1.41], Standard Error of Mean 1.112

50. Secondary Outcome: Absolute Values and Changes From Baseline in Fasting Plasma Glucose at at Days 2, 7, 14, 15, 21, 28 and 29 - Part A
Description: Fasting blood glucose samples were also collected on Days 0, 2, 7, and 15 for all cohorts, and on Days 21 and 29 for PF-06291874 100 mg Part A and PF-06291874 30 mg Part B.
Time Frame: predose on Days 0,2,7,14,15,21,28,29
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 18 | 12 | 12 | 12 | 14 | 12
mg/dL
  Baseline | 165.8 (31.61) | 163.6 (32.43) | 173.1 (38.28) | 173.9 (45.67) | 150.6 (29.45) | 170.4 (41.86)
  Day 2 absolute value: number analyzed (Participants) | 18 | 12 | 12 | 12 | 13 | 12
  Day 2 absolute value | 167.0 (35.06) | 158.7 (32.08) | 152.3 (31.59) | 150.0 (31.71) | 139.4 (42.05) | 135.1 (31.46)
  Day 2 changes from baseline: number analyzed (Participants) | 18 | 12 | 12 | 12 | 13 | 12
  Day 2 changes from baseline | 1.2 (16.60) | -4.9 (14.37) | -20.8 (13.54) | -23.9 (23.36) | -14.4 (32.29) | -35.3 (14.64)
  Day 7 absolute value: number analyzed (Participants) | 16 | 12 | 12 | 11 | 11 | 10
  Day 7 absolute value | 161.4 (33.30) | 154.5 (32.07) | 147.9 (27.04) | 138.5 (33.56) | 122.5 (16.38) | 116.5 (21.59)
  Day 7 changes from baseline: number analyzed (Participants) | 16 | 12 | 12 | 11 | 11 | 10
  Day 7 changes from baseline | -5.4 (18.14) | -9.1 (22.57) | -25.2 (25.83) | -37.4 (25.10) | -35.6 (21.67) | -38.4 (15.37)
  Day 14 absolute value | 150.9 (33.95) | 144.4 (33.67) | 133.3 (39.57) | 131.5 (28.68) | 112.9 (17.54) | 121.3 (30.03)
  Day 14 changes from baseline | -14.8 (29.96) | -19.2 (21.45) | -39.8 (34.07) | -42.4 (29.56) | -37.7 (19.46) | -49.1 (18.29)
  Day 15 absolute value: number analyzed (Participants) | 18 | 11 | 12 | 11 | 13 | 12
  Day 15 absolute value | 155.4 (33.08) | 150.9 (37.64) | 131.6 (25.96) | 132.7 (31.67) | 120.4 (22.15) | 122.7 (30.61)
  Day 15 changes from baseline: number analyzed (Participants) | 18 | 11 | 12 | 11 | 13 | 12
  Day 15 changes from baseline | -10.4 (27.51) | -16.2 (21.64) | -41.5 (33.08) | -44.2 (33.10) | -33.4 (24.46) | -47.7 (19.31)
  Day 21 absolute value: number analyzed (Participants) | 6 | 0 | 0 | 0 | 13 | 0
  Day 21 absolute value | 161.2 (38.22) |  |  |  | 128.5 (26.19) |
  Day 21 changes from baseline: number analyzed (Participants) | 6 | 0 | 0 | 0 | 13 | 0
  Day 21 changes from baseline | 1.1 (30.57) |  |  |  | -24.2 (31.40) |
  Day 28 absolute value: number analyzed (Participants) | 6 | 0 | 0 | 0 | 14 | 0
  Day 28 absolute value | 163.7 (26.90) |  |  |  | 122.4 (20.54) |
  Day 28 changes from baseline: number analyzed (Participants) | 6 | 0 | 0 | 0 | 14 | 0
  Day 28 changes from baseline | 3.6 (22.52) |  |  |  | -28.2 (15.99) |
  Day 29 absolute value: number analyzed (Participants) | 6 | 0 | 0 | 0 | 13 | 0
  Day 29 absolute value | 166.5 (31.56) |  |  |  | 129.6 (23.47) |
  Day 29 changes from baseline: number analyzed (Participants) | 6 | 0 | 0 | 0 | 13 | 0
  Day 29 changes from baseline | 6.4 (21.17) |  |  |  | -24.2 (21.52) |

51. Secondary Outcome: Absolute Values and Changes From Baseline in Fasting Plasma Glucose at Days 2, 7, 14, 15, 21, 28 and 29 - Part B
Description: as for outcome 50
Time Frame: Days 0,2,7,14,15,21,28,29
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 30 mg
Number analyzed (Participants) | 13 | 10 | 14
mg/dL
  Baseline | 156.0 (37.72) | 163.9 (31.43) | 154.3 (38.79)
  Day 2 absolute value: number analyzed (Participants) | 11 | 10 | 13
  Day 2 absolute value | 133.9 (26.73) | 147.6 (32.25) | 129.7 (28.13)
  Day 2 changes from baseline: number analyzed (Participants) | 11 | 10 | 13
  Day 2 changes from baseline | -11.8 (10.79) | -16.3 (9.05) | -29.7 (18.11)
  Day 7 absolute value: number analyzed (Participants) | 11 | 10 | 13
  Day 7 absolute value | 125.9 (32.13) | 134.4 (32.15) | 114.4 (20.67)
  Day 7 changes from baseline: number analyzed (Participants) | 11 | 10 | 13
  Day 7 changes from baseline | -23.0 (25.32) | -29.5 (15.47) | -41.6 (36.31)
  Day 14 absolute value: number analyzed (Participants) | 12 | 10 | 14
  Day 14 absolute value | 118.3 (40.08) | 128.6 (36.04) | 108.9 (24.64)
  Day 14 changes from baseline: number analyzed (Participants) | 12 | 10 | 14
  Day 14 changes from baseline | -31.0 (35.02) | -35.3 (18.32) | -45.3 (32.40)
  Day 15 absolute value: number analyzed (Participants) | 12 | 10 | 14
  Day 15 absolute value | 124.7 (37.44) | 133.4 (36.28) | 115.4 (32.53)
  Day 15 changes from baseline: number analyzed (Participants) | 12 | 10 | 14
  Day 15 changes from baseline | -24.6 (33.01) | -30.5 (19.31) | -38.8 (33.39)
  Day 21 absolute value: number analyzed (Participants) | 7 | 0 | 13
  Day 21 absolute value | 136.9 (34.54) |  | 131.5 (34.20)
  Day 21 changes from baseline: number analyzed (Participants) | 7 | 0 | 13
  Day 21 changes from baseline | -3.8 (26.23) |  | -18.3 (37.27)
  Day 28 absolute value: number analyzed (Participants) | 7 | 0 | 14
  Day 28 absolute value | 124.3 (21.84) |  | 113.3 (34.71)
  Day 28 changes from baseline: number analyzed (Participants) | 7 | 0 | 14
  Day 28 changes from baseline | -16.4 (33.19) |  | -41.0 (44.01)
  Day 29 absolute value: number analyzed (Participants) | 7 | 0 | 13
  Day 29 absolute value | 127.9 (15.87) |  | 127.5 (28.80)
  Day 29 changes from baseline: number analyzed (Participants) | 7 | 0 | 13
  Day 29 changes from baseline | -12.8 (11.53) |  | -26.1 (28.74)

52. Secondary Outcome: Absolute Values and Changes From Baseline in Fasting Plasma Insulin at Days 14 and 28 - Part A
Description: Fasting blood insulin samples were collected on Days -1, 14 and 28 for all cohorts, and on Day 28 for PF-06291874 100 mg Part A. Baseline was defined as the value on Day -1.
Time Frame: Days -1, 14, 28
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: µIU/mL
Arm/Group | Placebo | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 18 | 12 | 12 | 12 | 14 | 13
µIU/mL
  Baseline: number analyzed (Participants) | 18 | 12 | 12 | 12 | 14 | 12
  Baseline | 7.82 (3.26) | 9.84 (5.12) | 11.04 (6.06) | 7.34 (3.60) | 10.77 (6.62) | 9.64 (5.61)
  Day 14 absolute value: number analyzed (Participants) | 18 | 11 | 11 | 12 | 14 | 12
  Day 14 absolute value | 6.93 (3.91) | 9.83 (4.01) | 10.33 (4.96) | 5.61 (2.72) | 9.09 (4.27) | 8.98 (5.02)
  Day 14 changes from baseline: number analyzed (Participants) | 18 | 11 | 11 | 12 | 14 | 12
  Day 14 changes from baseline | -0.88 (2.81) | 0.00 (3.86) | -0.37 (3.46) | -1.73 (1.52) | -1.68 (3.43) | -0.66 (2.72)
  Day 28 absolute value: number analyzed (Participants) | 6 | 0 | 0 | 0 | 14 | 0
  Day 28 absolute value | 8.53 (4.20) |  |  |  | 9.30 (3.43) |
  Day 28 changes from baseline: number analyzed (Participants) | 6 | 0 | 0 | 0 | 14 | 0
  Day 28 changes from baseline | -0.82 (4.35) |  |  |  | -1.46 (3.20) |

53. Secondary Outcome: Absolute Values and Changes From Baseline in Fasting Plasma Insulin at Days 14 and 28 - Part B
Description: Fasting blood insulin samples were collected on Days -1, 14 and 28 for all cohorts, and on Day 28 for PF-06291874 30 mg Part B. Baseline was defined as the value on Day -1.
Time Frame: Days -1, 14, 28
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: µIU/mL
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 30 mg
Number analyzed (Participants) | 13 | 12 | 14
µIU/mL
  Baseline: number analyzed (Participants) | 13 | 9 | 14
  Baseline | 8.66 (2.59) | 14.49 (9.70) | 9.69 (4.94)
  Day 14 absolute value: number analyzed (Participants) | 11 | 10 | 12
  Day 14 absolute value | 8.08 (3.81) | 12.57 (8.63) | 9.82 (4.18)
  Day 14 changes from baseline: number analyzed (Participants) | 11 | 9 | 12
  Day 14 changes from baseline | -0.49 (2.96) | -1.13 (1.75) | -0.25 (4.07)
  Day 28 absolute value: number analyzed (Participants) | 7 | 0 | 13
  Day 28 absolute value | 7.96 (3.58) |  | 10.43 (4.50)
  Day 28 changes from baseline: number analyzed (Participants) | 7 | 0 | 13
  Day 28 changes from baseline | -0.44 (2.92) |  | 1.41 (4.52)

54. Secondary Outcome: Percent Change From Baseline in Lipid Parameters (mg/dL) by Treatment Group on Days 14 and 28 - Part A
Description: Blood samples (3.5 mL) for all lipids and 2 mL for ApoB100 were collected at Hour 0 Day 1, Day 7 prior to breakfast, Hour 0 Day 14 for all cohorts; Days 21 and 28 for PF-06291874 100 mg Part A and PF-06291874 30 mg Part B.
Time Frame: Days 0,14 and 28
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Placebo | PF-06291874 5 mg | PF-06291874 15 mg | PF-06291874 50 mg | PF-06291874 100 mg | PF-06291874 150 mg
Number analyzed (Participants) | 18 | 12 | 12 | 12 | 14 | 13
percentage of change
  Total Cholesterol-Day 14 Mean Percent Change | -8.6 (6.7) | -5.6 (6.6) | -5.6 (14.1) | 1.7 (11.8) | 0.0 (9.9) | 9.7 (10.3)
  Total Cholesterol-Day28 Mean Percent Change: number analyzed (Participants) | 6 | 0 | 0 | 0 | 14 | 0
  Total Cholesterol-Day28 Mean Percent Change | 1.4 (13.0) |  |  |  | 4.3 (13.3) |
  LDL Cholesterol -Day 14 Mean Percent Change | -9.6 (12.6) | -9.4 (10.8) | -6.4 (16.7) | 2.0 (17.9) | -0.4 (12.2) | 12.0 (18.3)
  LDL Cholesterol -Day28 Mean Percent Change: number analyzed (Participants) | 6 | 0 | 0 | 0 | 14 | 0
  LDL Cholesterol -Day28 Mean Percent Change | 1.8 (16.8) |  |  |  | 4.7 (14.0) |
  HDL Cholesterol -Day 14 Mean Percent Change | -5.4 (5.6) | -5.2 (11.3) | -6.5 (9.9) | -4.0 (9.7) | -1.5 (8.4) | 2.6 (12.7)
  HDL Cholesterol -Day28 Mean Percent Change: number analyzed (Participants) | 6 | 0 | 0 | 0 | 14 | 0
  HDL Cholesterol -Day28 Mean Percent Change | -4.3 (8.5) |  |  |  | 0.2 (10.7) |
  Triglycerides -Day 14 Mean Percent Change | -13.9 (15.2) | 6.4 (21.4) | 10.3 (30.5) | 11.6 (33.9) | -0.2 (23.9) | 18.3 (19.9)
  Triglycerides -Day28 Mean Percent Change: number analyzed (Participants) | 6 | 0 | 0 | 0 | 14 | 0
  Triglycerides -Day28 Mean Percent Change | 3.8 (24.5) |  |  |  | 6.4 (19.6) |
  ApoB100 -Day 14 Mean Percent Change | -7.2 (6.8) | -5.6 (9.9) | -6.1 (14.8) | 1.4 (10.8) | -0.2 (10.3) | 9.0 (11.0)
  ApoB100 -Day 28 Mean Percent Change: number analyzed (Participants) | 6 | 0 | 0 | 0 | 14 | 0
  ApoB100 -Day 28 Mean Percent Change | 0.7 (12.6) |  |  |  | 2.7 (10.0) |

55. Secondary Outcome: Percent Change From Baseline in Lipid Parameters (mg/dL) by Treatment Group on Days 14 and 28 - Part B
Description: as for outcome 54
Time Frame: Days 0,14 and 28
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 30 mg
Number analyzed (Participants) | 13 | 12 | 14
Percentage of change
  Total Cholesterol-Day 14 Mean Percent Change | -4.0 (12.6) | -0.6 (11.9) | -4.7 (8.4)
  Total Cholesterol-Day28 Mean Percent Change: number analyzed (Participants) | 6 | 0 | 14
  Total Cholesterol-Day28 Mean Percent Change | 8.4 (25.3) |  | -1.5 (7.7)
  LDL Cholesterol -Day 14 Mean Percent Change | -5.5 (15.6) | 1.50 (21.5) | -7.5 (14.2)
  LDL Cholesterol -Day28 Mean Percent Change: number analyzed (Participants) | 6 | 0 | 14
  LDL Cholesterol -Day28 Mean Percent Change | 15.7 (28.8) |  | -0.7 (10.0)
  HDL Cholesterol -Day 14 Mean Percent Change | -4.7 (12.9) | -5.8 (12.2) | -2.9 (10.6)
  HDL Cholesterol -Day28 Mean Percent Change: number analyzed (Participants) | 6 | 0 | 14
  HDL Cholesterol -Day28 Mean Percent Change | 7.8 (13.6) |  | 1.7 (11.2)
  Triglycerides -Day 14 Mean Percent Change | -18.6 (15.7) | -6.0 (17.5) | -8.4 (20.5)
  Triglycerides -Day28 Mean Percent Change: number analyzed (Participants) | 6 | 0 | 14
  Triglycerides -Day28 Mean Percent Change | 4.3 (60.9) |  | -1.9 (23.7)
  ApoB100 -Day 14 Mean Percent Change | -3.5 (12.4) | -4.1 (10.3) | -5.6 (10.7)
  ApoB100 -Day 28 Mean Percent Change: number analyzed (Participants) | 6 | 0 | 14
  ApoB100 -Day 28 Mean Percent Change | 12.7 (21.2) |  | -1.1 (4.5)

ADVERSE EVENTS:
Arm/Group | Part A: Placebo | Part A: PF-06291874 5 mg | Part A: PF-06291874 15 mg | Part A: PF-06291874 50 mg | Part A: PF-06291874 100 mg | Part A: PF-06291874 150 mg | Part B: Placebo | Part B: PF-06291874 15 mg | Part B: PF-06291874 30 mg | Total
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/12 | 0/12 | 0/12 | 0/14 | 0/12 | 0/13 | 0/10 | 0/14 | 0/117
Other Adverse Events (participants affected / at risk) | 10/18 | 7/12 | 4/12 | 6/12 | 5/14 | 3/12 | 8/13 | 5/10 | 5/14 | 53/117
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=18) | Part A: PF-06291874 5 mg (N=12) | Part A: PF-06291874 15 mg (N=12) | Part A: PF-06291874 50 mg (N=12) | Part A: PF-06291874 100 mg (N=14) | Part A: PF-06291874 150 mg (N=12) | Part B: Placebo (N=13) | Part B: PF-06291874 15 mg (N=10) | Part B: PF-06291874 30 mg (N=14) | Total (N=117)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chromatopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 7
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 9
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Application site bruise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 5
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 4
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 5
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 6
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 4
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.